CLINICAL TRIAL: NCT02756598
Title: Stress, Anxiety and Type A Personality and Analgesics. Impact on Induction Time and Consumption of Analgesics During Cardiac Surgery
Brief Title: Stress, Anxiety and Type A Personality and Analgesics
Acronym: SATA-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Carl-Johan Jakobsen, Consultant Anesthesiologist, Ass professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SATA-1
Record Dates: First submitted 2015-12-30; First posted 2016-04-29 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Postoperative; Dysfunction Following Cardiac Surgery
Keywords: sufentanil; propofol; personality/stress test; fast-track
MeSH Terms: interventions — Sufentanil; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sufentanil I (Active Comparator): Randomized arm "moderate" sufentanil I: bolus 1 microgram/kg propofol I: infusion 0.03 mg/kg/min
  Interventions: Drug: Sufentanil I; Drug: Propofol I
- Sufentanil II (Active Comparator): Randomized arm "low" sufentanil II bolus 0.5 microgram/kg propofol II: infusion 0.06 mg/kg/min
  Interventions: Drug: Sufentanil II; Drug: Propofol II

INTERVENTIONS:
Drug: Sufentanil I — bolus dose of sufentanil 1 microgram/kg
  Other Names: Sufenta
  Arms: Sufentanil I
Drug: Sufentanil II — bolus dose of sufentanil 0.5 microgram/kg
  Other Names: Sufenta
  Arms: Sufentanil II
Drug: Propofol I — Continued dose of propofol 0.03 mg/kg/min
  Other Names: Propofol
  Arms: Sufentanil I
Drug: Propofol II — Continued dose of propofol 0.06 mg/kg/min
  Other Names: Propofol
  Arms: Sufentanil II

SUMMARY:
Patients scheduled for elective cardiac surgery are preoperative evaluated using different personality type, stress and anxiety tests.

Patient are randomized to receive the investigators' standard moderate dose sufentanil (bolus 1microgram/kg and propofol 0.03 mg/kg/min) or low dose sufentanil (bolus 0.5 microgram/kg and propofol 0.06 mg/kg/min).

DETAILED DESCRIPTION:
Patients randomized and the type of induction informed to the anaesthetist 30 minutes before surgery.

Patients are monitored before induction of anesthesia. Propofol is started on the randomized infusion rate. Sufentanil bolus are given according to randomization. BIS level is followed. Time to reach BIS < 50 is monitored. BIS after 30, 60 and 90 minutes are registered. Lowest BIS during surgery are registered. Total amounts of sufentanil and propofol recorded.

ELIGIBILITY:
Inclusion Criteria:

* All elective cardiac surgery patients

Exclusion Criteria:

* Patients requiring special attention or monitoring during induction
* Patients with expected longer postoperative ventilation time
* Patients allergic to sufentanil and or propofol
* Participation in other projects
* Pregnancy

Ages: 16 Years to 90 Years | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Association between preoperative personality/stress/anxiety and time (minutes) to reach anaesthetic depth goal by bi-spectral index (BIS) | Up to 30 minutes
  Minutes to reach BIS 50
Potential of sufentanil regime on fast-track measured by ventilation time and association with eligible discharge from intensive care unit. | Up to 24 hours
  Postoperative ventilation time (hours/minutes) and the association to eligible discharge from ICU.

SECONDARY OUTCOMES:
Sufentanil regime and association to haemodynamic parameters (blood pressures, heart rate, cardiac output, oxygenation) | up to 24 hours
  Perioperative changes in haemodynamic parameters (analysis of varians) of haemodynamic parameters according to sufentanil regime
Association between preoperative personality/stress/anxiety tests and postoperative care using postoperative quality score | up to 24 hours
  Association of preoperative tests and the postoperative ICU quality scoring
Association between preoperative personality/stress/anxiety and total amounts of sufentanil and propofol | Up to 12 hours
  Amounts of drugs as pr kg pr time unit of involved drugs

IPD SHARING:
Plan to Share IPD: No